CLINICAL TRIAL: NCT06037954
Title: Mental Health Care Initiation Intervention for Older Adults With Cancer
Brief Title: A Study of Mental Health Care in People With Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 23-218
Record Dates: First submitted 2023-09-08; First posted 2023-09-14 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; Colorectal Cancer; Lung Cancer; Prostate Cancer
Keywords: 65 years and older; Mental health care; 23-218
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Lung Neoplasms; Prostatic Neoplasms | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Intervention Model Description: This protocol aims to refine and pilot test a brief telehealth intervention, Open Door for Cancer (OD-C), that addresses individual barriers to mental health service initiation in depressed older adults with cancer (OACs) without requiring in-person appointments.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open Door for Cancer (OD-C) (Experimental): OD-C includes five components delivered in three 30-minute telephone or videoconference visits over six weeks and one booster telephone call. All sessions are audio-recorded.
  Interventions: Other: 30-minute telephone or videoconference sessions
- Usual Care (Active Comparator): Participants assigned to Usual Care (n=50) will receive standard care. MSK's current usual care for distress screening is that all patients are screened for distress when they initiate care at MSK. Additional distress screening is conducted based on the determination of the oncology team. In addition, patients are referred to social work, psychology, and/or psychiatry based on the judgment of the oncology team.
  Interventions: Other: Questionnaires; Other: Interviews

INTERVENTIONS:
Other: Questionnaires — Patient demographic characteristics, Clinical variables, Cornell Service Index-Short Form (CSI), Patient Health Questionnaire-9 (PHQ-9), Generalized Anxiety Disorder scale-7 (GAD-7), Client Satisfaction Questionnaire (CSQ-8), Intention to Seek Help Scale, Health Beliefs about Mental Illness Instrument (HBMII) - Emotional/Nervous Severity Scale, Health Beliefs about Mental Illness Instrument (HBMII) - Emotional/Nervous Benefits Scale, Barriers to Mental Health Services Scale-Revised, Cues to action, Self-Efficacy to Seek Mental Health Care (SE-SMHC)
  Arms: Usual Care
Other: Interviews — Interviews will be conducted by the qualitative methods specialist and trained study staff and will last 30-45 minutes.
  Arms: Usual Care
Other: 30-minute telephone or videoconference sessions — Includes five components delivered in three 30-minute telephone or videoconference visits over six weeks and one booster telephone call. All sessions are audio-recorded. The five components are:
  1. Provide education about depression and treatment options
  2. Identify treatment preferences and a personal goal achievable with mental health care
  3. Assess barriers to treatment initiation
  4. Recommend a referral using standardized referral options
  5. Address barriers to accessing care
  Arms: Open Door for Cancer (OD-C)

SUMMARY:
The purpose of this study is to look at mental health services for adults with depressed mood who were diagnosed with cancer at the age of 65 or older. This study will compare the usual approach for connecting older adults with depressed mood to mental health services with the Open Door for Cancer (OD-C) approach. We will find out if the OD-C approach is practical and useful for cancer patients who participate in the intervention and for providers who see or treat cancer patients.

ELIGIBILITY:
Inclusion Criteria:

Patients

* Per medical record and/or self-report, diagnosed with breast, colorectal, lung, or prostate cancer at age 65 years or older
* Per medical record and/or self-report, undergoing active cancer treatment (e.g., radiation, chemotherapy, immunotherapy, surgery) or within six months of completing treatment
* Score of ≥5 on the Patient Health Questionnaire-9 (PHQ-9)
* Per self-report, fluent in English** ** Language verification: Prior to enrollment, patients will be asked the following two questions by a Clinical Research Coordinator (CRC) to verify English fluency necessary for participation in the study:

  1. How well do you speak English? (must respond "very well" or "well" when given the choices of Very well, Well, Not well, Not at all, Don't know, or Refused)
  2. What is your preferred language for healthcare? (must respond English)

Providers

* Per self-report, works in oncology, nursing, social work, psychology, or psychiatry
* Per self-report, currently works in oncology at least 50% of the time
* Per self-report, provided cancer care for at least three years at time of consent
* Per self-report, fluent in English

Exclusion Criteria:

Patients

* Severely cognitively impaired as demonstrated by Blessed Orientation Memory Concentration scores of ≥ 11
* Per research staff judgment and/or self-report, too ill or weak to complete study procedures
* Per medical record and/or self-report, receiving hospice care at the time of enrollment
* Per medical record and/or self-report, currently enrolled in mental health treatment

Providers

* N/A

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-09-07 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Refusal rates | 2 years
  ≥75% of eligible patients enroll in the study
Attrition rates | 2 years
  ≥80% of patients who enroll complete all study procedures

SECONDARY OUTCOMES:
Treatment satisfaction | 2 years
  Client Satisfaction Questionnaire-8 mean score of ≥3

CONTACTS AND LOCATIONS:
Overall Officials: Kelly McConnell, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm